CLINICAL TRIAL: NCT04340128
Title: Evaluation of Efficacy of Intra-lesional Injections of Glucantime Once Weekly in Comparison With Twice Weekly in the Treatment of Acute Anthroponotic Cutaneous Leishmaniasis (ACL)
Brief Title: Efficacy of Intra-lesional Injections of Glucantime Once a Week or Twice a Week in the Treatment of Anthroponotic Cutaneous Leishmaniasis (ACL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Mashad University of Medical Sciences (Unknown); Kerman University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: j/423/2252; 29463
Record Dates: First submitted 2011-02-16; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2011-02

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Anthroponotic Cutaneous Leishmaniasis; L. tropica; Meglumine antimoniate (Glucantime)
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate

ARMS (2):
- 1 (Active Comparator): Intra-lesional injection of Glucantime once a week
  Interventions: Drug: Meglumine antimoniate
- 2 (Experimental): Intra-lesional injection twice a week, 0.1/cm2
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Meglumine antimoniate — Intra-lesional injection once a week, 0.1/cm2
  Other Names: Glucantime
  Arms: 1
Drug: Meglumine antimoniate — Intra-lesional injection twice a week, 0.1/cm2
  Other Names: Glucantime
  Arms: 2

SUMMARY:
Anthroponotic Cutaneous Leishmaniasis (ACL) is a parasitic disease caused by Leishmania tropica, pentavalent antimonials (sodium stibogluconate and meglumine antimoniate) have been used as a standard treatment for leishmaniasis for last 80 years. Systemic antimonial injection is painful, toxic, not affordable and moreover is not always effective. Many different modalities are used to treat the disease with a limited success. Intra-lesional injections of antimonials are used for the treatment of patients with a few lesions but no data is available on the rate of efficacy. In this study the efficacy of intra-lesional injections of Glucantime weekly is compared with intra-lesional injections of Glucantime twice weekly.

ELIGIBILITY:
Inclusion Criteria:

* Parasitologically proven cases of CL based on positive smear and/or culture
* Otherwise healthy subjects on the basis of medical history.
* Age 9-70 years
* Willing to participate in the study and sign the informed consent (by the patient or his/her parent/guardian in case of younger than 18 years).

Exclusion Criteria:

* Pregnant or lactating women
* Duration of lesion more than 6 months
* Number of lesions more than 4
* History of allergy to Glucantime
* Serious systemic illnesses (as judged by the physician)
* Participation in any drug trials in the last 60 days
* No indication for systemic treatment

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Complete healing of the lesion(s) | 5 months

SECONDARY OUTCOMES:
Partiall cure | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Khatami, MD MSPH, Study Director — Center for Research & Training in Skin Diseases & Leprosy, Tehran University of Medical Sciences; Ali Khamesipour, PhD, Principal Investigator — Center for Research & Training in Skin Diseases & Leprosy, Tehran University of Medical Sciences; Mahdieh Bahrami, MD, Study Chair — Kerman University of Medical Sciences; Mohammad Hossein Ghoorchi, MD, Study Chair — Mashhad University of Medical Sciences
Locations (1):
- CRTSDL, Tehran, Iran